CLINICAL TRIAL: NCT03609697
Title: Effects of a Community-based Weight Loss Programme Targetting Chinese Overweight Adults With Pre-diabetes: A Randomized Controlled Trial
Brief Title: A Community-based Weight Loss Programme for Chinese Overweight Adults With Pre-diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Mandy M. Ho, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HCPS01170498
Record Dates: First submitted 2018-07-13; First posted 2018-08-01 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Pre-diabetes
Keywords: Diabetes prevention; Pre-diabetes; Weight loss; Cardio-metabolic risks; Obesity; Lifestyle intervention; Community-based
MeSH Terms: conditions — Glucose Intolerance; Weight Loss; Obesity

STUDY DESIGN:
Intervention Model Description: It is a 12-month 2-arm randomised controlled trial, RCT (the lifestyle intervention group and the SMS intervention group) with a 3 year follow up. The programme will proceed in two phases: the intensive intervention phase (0-6 months) and the maintenance phase (7-12 months). During the intensive intervention phase, participants in the lifestyle intervention group will attend 7 group-based interventions plus two sessions of individual face-to-face dietician consultation. During the maintenance phase, participants will receive monthly phone call from the research team.
  The SMS intervention group will receive regular SMS during both the intensive intervention and the maintenance phases.
Who Masked: Outcomes Assessor
Masking Description: All outcome assessors will be blinded to group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community-based lifestyle intervention (Experimental): Participants will attend 7 community-based group intervention sessions plus 2 individual face-to-face dietician consultation sessions during the first 6 months, followed by a 6-month maintenance phase which they will receive monthly phone support from the research team.
  Interventions: Behavioral: group-based lifestyle intervention
- Minimal intervention (SMS intervention) (Other): Participants will receive one SMS per month during the first 6 months, followed by a 6-month maintenance phase which participants will receive one SMS every 2 months.
  Interventions: Behavioral: Minimal intervention (SMS intervention)

INTERVENTIONS:
Behavioral: group-based lifestyle intervention — Involve education about pre-diabetes self-management, weight loss, behavioural modification skills, nutrition and physical activity.
  Other Names: individual dietitian consultation; Telephone support; community-based intervention
  Arms: Community-based lifestyle intervention
Behavioral: Minimal intervention (SMS intervention) — Text message related to general information about T2DM, pre-diabetes, and lifestyle modification.
  Arms: Minimal intervention (SMS intervention)

SUMMARY:
Type 2 diabetes (T2DM) is a serious chronic condition and one of the world's fastest growing health problems. The onset of T2DM is gradual, with most individuals progressing through a state of pre-diabetes. Pre-diabetes is a prevalent and potentially reversible condition, which provides an important window of opportunity for the prevention of T2DM and its complications. This project aims to translate the evidence-based diabetes prevention strategies into a community setting to reduce diabetes risks in Hong Kong Chinese people with pre-diabetes .

DETAILED DESCRIPTION:
Type 2 diabetes (T2DM) is a major non-communicable disease and one of the world's fastest growing health problem. It is associated with significant morbidity, including increased risk of heart disease and stroke, hypertension, retinopathy and blindness, renal failure and leg amputation, which place an enormous burden on individuals, society and the healthcare system. The T2DM trend in Hong Kong mirrors the global trend. It is a major cause of mortality and morbidity with approximately 700,000 people diagnosed with diabetes, representing 10% of Hong Kong's total population.

T2DM is a non-reversible, yet a preventable condition. The onset of T2DM is gradual, with most individuals progressing through a state of pre-diabetes. People with pre-diabetes, defined as having impaired fasting glucose (IFG), impaired glucose tolerance (IGT) or elevated glycated haemoglobulin (HbA1C) , are at increased risk of developing T2DM and its associated complications, such as heart diseases and retinopathy, which can develop even in the absence of progression to overt T2DM. Hence, it is essential that people with pre-diabetes are targeted for early intervention to prevent T2DM and related complications.

International clinical trials demonstrated that lifestyle interventions targeting at least 5% weight loss in individuals with pre-diabetes can be cost-effective in preventing T2DM. Lifestyle intervention (which includes diet, physical activity and behavioural modification components) and self-management of pre-diabetes has been listed as an effective means of decreasing the incidence of T2DM in the international guidelines on management of pre-diabetes.

The aim of this study is to translate preventive research into effective community-based intervention by setting up a culturally appropriate lifestyle intervention programme for the prevention of T2DM in Hong Kong Chinese adults with pre-diabetes.

ELIGIBILITY:
Inclusion Criteria:

* aged 30 to 65 years
* overweight (BMI ≥ 23kg/m2) or obese (BMI ≥ 25 kg/m2)
* with at least one blood test result showing IGT (7.8-11.0 mmol/L after a two-hour glucose tolerance test), IFG (fasting glucose 5.6 - 6.9 mmol/L) or impaired HbA1c 5.7% - 6.4%
* have a mobile phone
* able to read Chinese and speak Cantonese.

Exclusion Criteria:

* with current or clinical history of T2DM, or with co-morbid conditions that may limit participation in the study, such as recent history of an acute cardiovascular event, uncontrolled hypertension, cancer or major psychiatric or cognitive problems
* already participating in a weight loss programme
* receiving drug treatment for pre-diabetes (e.g. Metformin) or long-term use of medications known to influence glucose metabolism (e.g. corticosteroids)

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2018-08-10 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Percent weight change | % weight change from baseline at 6-month and 12-months
  % weight change from baseline

SECONDARY OUTCOMES:
Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) | Changes from baseline insulin sensitivity at 6-month and 12-months
  Estimated from fasting insulin and fasting glucose, [fasting insulin (uU/mL)*fasting glucose(mmol/L)]/22.5
Fasting insulin | Changes from baseline fasting insulin at 6-month and 12-months
  Fasting insulin
Fasting blood glucose (FG) | Changes from baseline FG at 6-month and 12-months
  Fasting blood glucose
Haemoglobin A1C (HbA1C) | Changes from baseline HbA1Cat 6-month and 12-months
  HbA1C
Systolic and diastolic blood pressure (SBP, DBP) | Changes from baseline SBP and DBP at 6-month and 12-months
  measured by automatic BP monitor
Blood lipid profile | Changes from baseline blood lipid to 6-month and 12-months
  fasting blood for total cholesterol, HDL, LDL and triglycerides
Diabetes status | 6-month and 12-months follow-up
  Oral glucose tolerance test
Physical activity | Change in levels of physical activity from baseline to 6-month and 12-months
  International physical activity questionnaire short form (IPAQ, Chinese version). A validated 6-item questionnaire to assess the frequency and duration of vigorous intensity activity, moderate intensity activity, and walking. The questionnaire will be scored using established methods (www.ipaq.ki.se). Data will be summarized to report physical activity in categories:
  1. High-active group
     * Vigorous-intensity activity on ≥ 3 days and accumulating ≥1500 MET-minutes/week OR
     * ≥7 days of any combination of walking, moderate-intensity or vigorous intensity activities achieving ≥3000 MET-minutes/week
  2. Moderate-active group
     * ≥3 days of vigorous activity of ≥20 minutes/day OR
     * ≥5 days of moderate-intensity activity or walking of ≥30 minutes/day OR
     * ≥5 days of any combination of walking, moderate-intensity or vigorous intensity activities achieving ≥600 MET-min/week.
  3. Low-active/inactive group Individuals who do not meet criteria for high- and moderate-active
Dietary intake | Changes in dietary intake from baseline to 6-month and 12-months
  24 hour recalls
Health-related quality of life (HRQOL) | Changes in HRQOL from baseline to 6-month and 12-months
  12-item Short Form Survey (SF12 Chinese version). It is a validated scale which provides two summary measures. Physical and Mental Health Composite Scores (PCS & MCS) will be computed using the scores of 12 questions and range from 0 to 100. Higher scores represent better health.
Carotid artery intima-media thickness (cIMT) | Change in cIMT from baseline to 6-month and 12-months
  High-resolution B-mode ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Dr Mandy Ho, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.

REFERENCES:
- [Background] Guariguata L, Whiting DR, Hambleton I, Beagley J, Linnenkamp U, Shaw JE. Global estimates of diabetes prevalence for 2013 and projections for 2035. Diabetes Res Clin Pract. 2014 Feb;103(2):137-49. doi: 10.1016/j.diabres.2013.11.002. Epub 2013 Dec 1. PMID 24630390
- [Background] American Diabetes Association. (2) Classification and diagnosis of diabetes. Diabetes Care. 2015 Jan;38 Suppl:S8-S16. doi: 10.2337/dc15-S005. No abstract available. PMID 25537714
- [Background] Yoon KH, Lee JH, Kim JW, Cho JH, Choi YH, Ko SH, Zimmet P, Son HY. Epidemic obesity and type 2 diabetes in Asia. Lancet. 2006 Nov 11;368(9548):1681-8. doi: 10.1016/S0140-6736(06)69703-1. PMID 17098087
- [Background] Hospital Authority of Hong Kong. Hospital Authority Statistical Report 2009-2010 [Internet]. Hong Kong; 2011 [cited 2015 Jan 26 ]. 182 p. Available from: http://www.ha.org.hk/ho/corpcomm/Statistical%20Report/2009-10.pdf
- [Background] Levitan EB, Song Y, Ford ES, Liu S. Is nondiabetic hyperglycemia a risk factor for cardiovascular disease? A meta-analysis of prospective studies. Arch Intern Med. 2004 Oct 25;164(19):2147-55. doi: 10.1001/archinte.164.19.2147. PMID 15505129
- [Background] Nathan DM, Davidson MB, DeFronzo RA, Heine RJ, Henry RR, Pratley R, Zinman B; American Diabetes Association. Impaired fasting glucose and impaired glucose tolerance: implications for care. Diabetes Care. 2007 Mar;30(3):753-9. doi: 10.2337/dc07-9920. No abstract available. PMID 17327355
- [Background] Singleton JR, Smith AG, Russell JW, Feldman EL. Microvascular complications of impaired glucose tolerance. Diabetes. 2003 Dec;52(12):2867-73. doi: 10.2337/diabetes.52.12.2867. PMID 14633845
- [Background] Pan XR, Li GW, Hu YH, Wang JX, Yang WY, An ZX, Hu ZX, Lin J, Xiao JZ, Cao HB, Liu PA, Jiang XG, Jiang YY, Wang JP, Zheng H, Zhang H, Bennett PH, Howard BV. Effects of diet and exercise in preventing NIDDM in people with impaired glucose tolerance. The Da Qing IGT and Diabetes Study. Diabetes Care. 1997 Apr;20(4):537-44. doi: 10.2337/diacare.20.4.537. PMID 9096977
- [Background] Ramachandran A, Snehalatha C, Mary S, Mukesh B, Bhaskar AD, Vijay V; Indian Diabetes Prevention Programme (IDPP). The Indian Diabetes Prevention Programme shows that lifestyle modification and metformin prevent type 2 diabetes in Asian Indian subjects with impaired glucose tolerance (IDPP-1). Diabetologia. 2006 Feb;49(2):289-97. doi: 10.1007/s00125-005-0097-z. Epub 2006 Jan 4. PMID 16391903
- [Background] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527
- [Background] Gong Q, Gregg EW, Wang J, An Y, Zhang P, Yang W, Li H, Li H, Jiang Y, Shuai Y, Zhang B, Zhang J, Gerzoff RB, Roglic G, Hu Y, Li G, Bennett PH. Long-term effects of a randomised trial of a 6-year lifestyle intervention in impaired glucose tolerance on diabetes-related microvascular complications: the China Da Qing Diabetes Prevention Outcome Study. Diabetologia. 2011 Feb;54(2):300-7. doi: 10.1007/s00125-010-1948-9. Epub 2010 Nov 3. PMID 21046360
- [Background] Lindstrom J, Peltonen M, Eriksson JG, Ilanne-Parikka P, Aunola S, Keinanen-Kiukaanniemi S, Uusitupa M, Tuomilehto J; Finnish Diabetes Prevention Study (DPS). Improved lifestyle and decreased diabetes risk over 13 years: long-term follow-up of the randomised Finnish Diabetes Prevention Study (DPS). Diabetologia. 2013 Feb;56(2):284-93. doi: 10.1007/s00125-012-2752-5. Epub 2012 Oct 24. PMID 23093136
- [Background] Twigg SM, Kamp MC, Davis TM, Neylon EK, Flack JR; Australian Diabetes Society; Australian Diabetes Educators Association. Prediabetes: a position statement from the Australian Diabetes Society and Australian Diabetes Educators Association. Med J Aust. 2007 May 7;186(9):461-5. doi: 10.5694/j.1326-5377.2007.tb00998.x. PMID 17484708
- [Background] Payne WR, Walsh KJ, Harvey JT, Livy MF, McKenzie KJ, Donaldson A, Atkinson MG, Keogh JB, Moss RS, Dunstan DW, Hubbard WA. Effect of a low-resource-intensive lifestyle modification program incorporating gymnasium-based and home-based resistance training on type 2 diabetes risk in Australian adults. Diabetes Care. 2008 Dec;31(12):2244-50. doi: 10.2337/dc08-0152. Epub 2008 Sep 16. PMID 18796621
- [Background] Katula JA, Vitolins MZ, Rosenberger EL, Blackwell CS, Morgan TM, Lawlor MS, Goff DC Jr. One-year results of a community-based translation of the Diabetes Prevention Program: Healthy-Living Partnerships to Prevent Diabetes (HELP PD) Project. Diabetes Care. 2011 Jul;34(7):1451-7. doi: 10.2337/dc10-2115. Epub 2011 May 18. PMID 21593290
- [Derived] Ho M, Chau PH, Yu EYT, Ying MT, Lam CLK. Community-based weight loss programme targeting overweight Chinese adults with pre-diabetes: study protocol of a randomised controlled trial. BMJ Open. 2020 Apr 8;10(4):e035196. doi: 10.1136/bmjopen-2019-035196. PMID 32273317